CLINICAL TRIAL: NCT03360721
Title: A Phase 2, Study of Apalutamide and Abiraterone Acetate in Castration-Resistant Metastatic Prostate Cancer Patients Evaluating a Predetermined Biomarker Signature
Brief Title: Apalutamide, Abiraterone Acetate, and Prednisone in Treating Participants With Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0060; NCI-2018-01054 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0060 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Castration-Resistant Prostate Carcinoma; Prostate Adenocarcinoma Without Neuroendocrine Differentiation; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (abiraterone acetate, apalutamide, prednisone) (Experimental): Participants receive abiraterone acetate PO once daily QD, apalutamide PO QD, and prednisone PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Yonsa; Zytiga
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; Erleada; JNJ 56021927; JNJ-56021927
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies how well apalutamide and abiraterone acetate work in treating participants with castration resistant prostate cancer that has spread to other places in the body (metastatic). Abiraterone acetate and apalutamide may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunosuppressive therapy, such as prednisone, is used to decrease the body's immune response and may improve bone marrow function. Giving apalutamide, abiraterone acetate, and prednisone may work better in treating participants with castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the radiographic progression free survival (PFS) of men with metastatic castration resistant prostate cancer (mCRPC) who are selected for treatment based on positive biomarker signature.

SECONDARY OBJECTIVES:

I. Safety. II. Composite progression free survival (PFSc) defined by Prostate Cancer Working Group 2 (PCWG2) (radiographic progression, prostate specific antigen [PSA] progression, or clinical deterioration).

III. Overall survival. IV. Exploratory biomarker analyses. V. Measures of prostate specific antigen (PSA) decline and associations with outcome.

VI. Radiologic response by PCWG2 criteria. VII. Measures of circulating tumor cell (CTC) and conversion to undetectable and/or favorable < 5.

OUTLINE:

Participants receive abiraterone acetate orally (PO) once daily (QD), apalutamide PO QD, and prednisone PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up for up to 16 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Presence of metastatic disease that can be biopsied by any methodology applicable
* Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., surgical or medical castration)
* Serum testosterone level =< 50 ng/dL at the screening visit
* Progressive disease defined as one or more of the following three criteria (NOTE: Patients who received an antiandrogen must demonstrate disease progression following discontinuation of antiandrogen):

  * PSA progression defined by a minimum of two rising PSA levels with an interval of >= 1 weeks between each determination. The PSA value at the screening visit should be >= 2 ng/mL
  * Soft tissue disease progression as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
  * Bone disease progression defined by two or more new lesions on bone scan
* Patients previously treated with chemotherapy must have no more than two prior chemotherapy regimens for the treatment of metastatic prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Serum albumin >= 3.0 g/dL
* Serum potassium >= 3.5 mmol/L
* Estimated life expectancy of >= 6 months
* Able to swallow the study drug and comply with study requirements
* Willing and able to give informed consent
* Tumor specimen obtained prior to treatment initiation by interventional radiology guided biopsy will be interrogated per immunohistochemistry (IHC) and features should be as follows for a patient to be eligible

  * Overexpression of androgen receptor (AR)-C terminal and AR-N terminal and PTEN with lack of ARV7 expression along with and ki67 =<10%
  * No combined RB loss and p53 mutation and
  * No expression of neuroendocrine markers CD56 and chromogranin (all markers assessed by standardized IHC protocols)
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. Must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug

  * The methods must consist of a condom and the use of another barrier method (such as a diaphragm or cervical/vault caps) with a spermicidal agent. Your female partner can choose to use an intrauterine device or system (intrauterine device [IUD] or intrauterine system [IUS]) or use birth control pills, injections, or implants instead of a barrier method

Exclusion Criteria:

* Known allergy to the study drugs or any of its components
* Severe, concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Known metastases to the brain
* Absolute neutrophil count < 1000/uL at the screening visit
* Platelet count =< 100,000 x 10^9/uL at the screening visit
* Hemoglobin < 9 g/dL at the screening visit at the screening visit
* NOTE: patients may not have received any growth factors or blood transfusions within seven days of the hematologic laboratory values obtained at the screening visit
* Total bilirubin (Tbili) > 1.5 times the upper limit of normal at the screening visit
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at the screening visit
* Creatinine (Cr) > 2 mg/dL at the screening visit
* History of another malignancy within the previous 2 years with > 30 % probability of relapse other than curatively treated non-melanomatous skin cancer
* Treatment with androgen receptor antagonists (bicalutamide, flutamide, nilutamide), 5-alpha reductase inhibitors (finasteride, dutasteride), estrogens, chemotherapy, or biologic therapy within 4 weeks of enrollment (day 1 visit)
* Radiation therapy within 3 weeks (if single fraction of radiotherapy within 2 weeks) of enrollment (day 1 visit)
* Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
* Structurally unstable bone lesions suggesting impending fracture
* History of seizure or any condition that may increase the patient's seizure risk. Also, history of loss of consciousness or transient ischemic attack within 12 months of day 1
* Clinically significant cardiovascular disease including:

  * Myocardial infarction within 6 months
  * Uncontrolled angina within 6 months
  * Congestive heart failure New York Heart Association (NYHA) class 3 or 4 in the past, or history of anthracycline or anthracenedione (mitoxantrone) treatment, unless a screening echocardiogram or multi-gated acquisition scan (MUGA) performed within three months results in a left ventricular ejection fraction that is >= 45%
  * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
  * Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on the screening electrocardiogram (ECG) > 470 msec
  * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
  * Hypotension (systolic blood pressure < 86 millimeters of mercury or bradycardia with a heart rate of < 50 beats per minute on any ECG taken at the screening visit
  * Bradycardia with a heat rate of < 50 beats per minutes in the screening ECG, unless pharmaceutically induced and reversible
  * Chronically uncontrolled hypertension as indicated by consistently elevated resting blood pressure (systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg) during screening
* Have used or plan to use from 30 days prior to enrollment (day 1 visit) through the end of the study the following medications known to lower the seizure threshold:

  * Aminophylline/theophylline
  * Atypical antipsychotics (e.g., clozapine, olanzapine, risperidone, ziprasidone)
  * Bupropion
  * Insulin
  * Lithium
  * Pethidine
  * Phenothiazine antipsychotics (e.g., prochlorperazine [compazine], chlorpromazine, mesoridazine, thioridazine)
  * Tricyclic and tetracyclic antidepressants (e.g., amitriptyline, desipramine, doxepin, imipramine, maprotiline, mirtazapine)
* Prior use of ketoconazloe, enzalutamide, abiraterone or apalutamide or participation in a previous clinical trial of ketoconazloe,enzalutamide, abiraterone or apalutamide unless within the neoadjuvant setting
* Use of an investigational agent within 4 weeks of enrollment (day 1)
* Gastrointestinal disorder affecting absorption (e.g., gastrectomy)
* Major surgery within 4 weeks prior to enrollment (day 1)
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's' disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * History of gastrointestinal (GI) bleeding within one year
* Known active or symptomatic viral hepatitis or chronic liver disease
* Known history of pituitary or adrenal dysfunction
* Baseline moderate and severe hepatic impairment (Child Pugh class B & C)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From enrollment until radiographic progression, death from any cause, start of other therapy or last follow-up without progression, whichever comes first assessed up to 28 months
  Will be assessed using primary analysis set (PAS). Kaplan-Meier curves will be presented.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 28 months
  Will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 with grade and attribution to study drug.
Composite progression free survival (PFSc) | From protocol treatment start until Prostate Cancer Working Group 2 (PCWG2) progression (radiographic progression, PSA progression, or clinical deterioration), death, starting new treatment or last follow-up without PCWG2 progression
  Will be assessed using PAS.
Overall survival (OS) | Baseline until death or last contact, assessed up to 28 months
  Will be assessed using PAS.
Androgen expression signaling | Baseline to week 13
  Will be assessed using marker evaluable set (MES). The association between the biomarker and PSA level will be estimated using Spearman's rank correlation.
Survival escape pathway signaling | Baseline to week 13
  Will be assessed using MES.
PSA measurement | Up to 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Bagi Jana, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org